CLINICAL TRIAL: NCT03537885
Title: Development of an EEG Analytics Tool to Determine Effectiveness of a tDCS Protocol
Brief Title: EEG Analytics to Determine Effectiveness of a tDCS Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burke Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BRC493
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Healthy; EEG; Transcranial Magnetic Stimulation
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TMS, EEG, and tDCS Group (Experimental): Participants will wear a cap fitted with Electroencephalography (EEG) electrodes to detect the brain's activity during the task. Transcranial Magnetic Stimulation will be used to evaluate the brain's responsiveness to Transcranial Direct Current Stimulation.
  All study participants will receive the same study procedures - TMS, tDCS, and EEG.
  Interventions: Diagnostic Test: Transcranial Direct Current Stimulation; Diagnostic Test: Transcranial Magnetic Stimulation; Diagnostic Test: Electroencephalography (EEG)

INTERVENTIONS:
Diagnostic Test: Transcranial Direct Current Stimulation — Electrodes are placed on that head to deliver a non-invasive brain stimulation to the target area.
Diagnostic Test: Transcranial Magnetic Stimulation — A coil is held tangential to the head in order to deliver a non-invasive brain stimulation to the target area.
Diagnostic Test: Electroencephalography (EEG) — A cap is placed on the head with sensors to detect brain activity during the intervention.

SUMMARY:
The goal of this study is to monitor the brain using electroencephalography (EEG) while transcranial direct current stimulation (tDCS) is being administered, as a potential pathway to determine neurophysiological markers capable of forecasting the intensity of a subject's response to tDCS.

DETAILED DESCRIPTION:
Transcranial direct current stimulation is a non-invasive neuromodulation technique that has been the subject of many recent investigations. There is a growing body of evidence to suggest that tDCS can enhance the efficacy of various therapies. However, progress in the field is slow: many studies suffer from reproducibility issues, or highly variable results, including stroke rehabilitation. It is feasible that much of the variance in experimental results can be explained by an inability to quantitatively track individual responses to tDCS in real-time, and personalize stimulation parameters for maximum effect.

Monitoring the brain via EEG while tDCS is being administered is a potential pathway to determine neurophysiological markers capable of forecasting the intensity of a subject's response to tDCS. This research has not previously been attempted due to technical difficulties- namely, the electromagnetic interference that is associated with tDCS degrades EEG signal quality. Recent advances in electrode and amplification technology have made it possible to make EEG recordings simultaneously with tDCS.

The investigators will attempt to determine whether specific EEG signatures can indicate the magnitude of a tDCS response. Subjects will receive either real or sham anodal tDCS to the hand representation of their left primary motor cortex.

The efficacy of the tDCS protocol will be quantitatively determined using transcranial magnetic stimulation (TMS) to generate a motor-evoked potential (MEP) in the hand pre- and post-tDCS. Additionally, prior to, during, and following the tDCS protocol, we will record EEG event-related potentials (ERPs) in response to a finger-tapping (motor) task.

The investigators aim to draw a correlation between the magnitude of MEP changes and pre- and post-tDCS and changes in recorded ERPs before, during and after tDCS in order to quantify the response to tDCS over the motor cortex. If EEG metrics can be used to gauge efficacy in real-time during tDCS administration, the investigators will gain significant insight into how to appropriately and quantitatively individualize tDCS dosage parameters for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Neurologically healthy

Exclusion Criteria:

* Ongoing use of CNS-active medications
* Ongoing use of psychoactive medications, such as stimulants, antidepressants, and anti-psychotic medications
* Presence of a potential tDCS/TMS Risk Factor:

  1. Damaged skin at the site of stimulation (i.e. skin with ingrown hairs, acne, razor nicks, wounds that have not healed, recent scar tissue, broken skin, etc)
  2. Presence of an electrically, magnetically or mechanically activated implant (including cardiac pacemaker), an intracerebral vascular clip or any other electrically sensitive support system
  3. Metal in any part of the body, including metal injury to the eye (Jewelry must be removed during stimulation)
  4. A history of medication-resistant epilepsy in the family
  5. Past history of seizures or unexplained spells of loss of consciousness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Motor Evoked Potential | Within session
  A measure of the muscle's responsiveness to non-invasive stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Burke Medical Research Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers at this time.